CLINICAL TRIAL: NCT00499837
Title: Double-Blind, Randomized, Placebo-Controlled, Phase II Study of the Safety and Efficacy of Inhaled Alpha-1 Antitrypsin (AAT ) in Cystic Fibrosis Patients
Brief Title: Phase II Study of the Safety and Efficacy of Inhaled Alpha-1 Antitrypsin (AAT ) in Cystic Fibrosis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kamada, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Kamada-AAT (inhaled)-003
Record Dates: First submitted 2007-07-11; First posted 2007-07-12 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-04

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 80 mg/kg AAT inhaled (Experimental): 80 mg/kg AAT inhaled
  Interventions: Drug: Aerosolized, human, plasma-derived Alpha-1 Antitrypsin
- Placebo inhaled (Placebo Comparator): Placebo inhaled
  Interventions: Drug: Aerosolized, human, plasma-derived Alpha-1 Antitrypsin

INTERVENTIONS:
Drug: Aerosolized, human, plasma-derived Alpha-1 Antitrypsin

SUMMARY:
Cystic Fibrosis (CF) is an inherited disorder in which mucus-secreting glands in the lungs produce considerable quantity of thick, sticky secretions that clog the airways, promote bacterial growth and lead to chronic obstruction, inflammation and destruction of the airways.

The purpose of this study is to collect data about the resolution of the chronic inflammatory state in addition to assure the safety of the therapy in CF patients.

DETAILED DESCRIPTION:
In CF patients the unregulated inflammatory response overwhelms the normal protease (elastase)/antiprotease (AAT) balance, leading to the accumulation of elastase in the lung, destruction of the lung architecture, severe pulmonary dysfunction, and ultimately death.

Administration of AAT is to address the elastase/antiprotease imbalance in order to prevent destruction of the lung tissue and reduce the inflammatory dysregulation that causes pulmonary dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CF by clinical symptoms and positive sweat test or disease inducing mutation.
* Age >5 yrs
* Proven ability to perform reproducible PFTs
* FEV1 >25% predicted
* Steady disease state for 3 months and no decrease in lung function exceeding 10% during that period
* Colonization
* Stable concomitant therapy >2 weeks prior to visit 1 and during the study
* Non-tobacco user of any kind
* Ability for sputum induction
* Written informed consent

Exclusion Criteria:

* Severe CF with an FEV1 of <25% predicted
* History of lung transplant
* Active allergic bronchopulmonary aspergillosis (ABPA)
* Treatment with additional antibiotics (beyond standard CF treatment) for a period of 14 days before study entry (routine antibiotics permitted)
* Treatment with additional oral and/or IV steroids (beyond standard CF treatment) for a period of 14 days before study entry (screening day)
* Known hypersensitivity to plasma products
* IgA deficiency
* Uncontrolled hypertension
* Lung surgery in the previous two years
* Being on any thoracic surgery waiting list
* Severe concomitant disease
* Hospitalization within 1 month before study entry, not due to an airway disease
* Severe liver cirrhosis with ascites
* Hypersplenism
* Grade III/IV oesophageal varices
* Active pulmonary exacerbation within the 4 weeks prior to screening
* History of significant hemoptysis within the previous year
* Use of tobacco products or recreational drugs
* Pregnancy or breastfeeding
* Any serious or active medical or psychiatric illness which, in the opinion of the investigator, would interfere with patient treatment, assessment, or compliance with the protocol.
* Being a female of child-bearing age without adequate contraception
* Participation in research study within 1 month

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-09; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Safety and airway inflammation | days 1,7,14,21,28,35,42,49,56,63

SECONDARY OUTCOMES:
Sputum microbiology, pulmonary function and serum CRP | days 1,7,14,21,28,35,42,49,56,63

CONTACTS AND LOCATIONS:
Overall Officials: Eitan Kerem, MD, Principal Investigator — Hadassah Hebrew University, Medical Center, Mt. Scopus, Jerusalem
Locations (1):
- Hadassah Hebrew University, Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No